CLINICAL TRIAL: NCT03744884
Title: Movement Impairment Characterization and Rehabilitation for Spastic/Dystonic Cerebral Palsy Using Robotic Haptic Feedback in Virtual Reality
Brief Title: Movement Characterization in Spastic/Dystonic Cerebral Palsy Using Haptic Feedback in Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: OSF Healthcare System (Other); University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Principal Investigator, Citlali Lopez-Ortiz, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18476
Record Dates: First submitted 2018-10-26; First posted 2018-11-16 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Cerebral Palsy, Mixed; Cerebral Palsy, Spastic
Keywords: Virtual reality; Haptic feedback; Robotic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A group of children with dystonic or spastic/dystonic cerebral palsy and a group of typical developing children will be randomly assigned to an intervention or control group. The control group will only attend assessment sessions whereas the intervention group will attend both the assessment and intervention sessions.
Who Masked: Outcomes Assessor
Masking Description: Research team members administering clinical assessments will be blinded from participant allocation. Participant's allocation will not be revealed during the course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CP intervention group (Experimental): Force efforts with haptic feedback in virtual reality for participants with CP.
  Interventions: Behavioral: Force efforts with haptic feedback in virtual reality.
- CP control group (No Intervention): Regular activity control group, for participants with CP.
- TD intervention group (Experimental): Force efforts haptic feedback in virtual reality. The intervention will be the same as the CP intervention group but for typically developing participants.
  Interventions: Behavioral: Force efforts with haptic feedback in virtual reality.
- TD control group (No Intervention): Regular activity control group, same as CP no intervention group, but for typically developing participants.

INTERVENTIONS:
Behavioral: Force efforts with haptic feedback in virtual reality. — A virtual reality game-based intervention incorporating fully-automated robotic haptic feedback. The study consists of face-to-face assessments of movement before, after, and one-month following the completion of the six-session game-based intervention. Children with spastic/dystonic cerebral palsy between the ages of 7 and 17 will be recruited for this study along with a group of typically developing children in the same age range. Both groups of children will be randomly allocated into an intervention or control group using a blocked randomization method.
  Arms: CP intervention group; TD intervention group

SUMMARY:
This game-like intervention using virtual reality will provide an objective and quantitative characterization of dystonia and spasticity presentations in cerebral palsy, even if combined, through the process of motor learning. This intervention could have a therapeutic benefit in the rehabilitation of children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is the most common developmental motor disorder in children. Individuals with cerebral palsy demonstrate abnormal muscle tone and motor control. Within the population of children with cerebral palsy, between 4% and 17% present dystonic symptoms and between 80% to 95% of cases present spasticity. In many cases spasticity and dystonia are present in the same child and accurate diagnosis may be challenging.

This study consists of a randomized controlled trial that uses a virtual reality game-based intervention incorporating fully-automated robotic haptic feedback to aid the the objective, quantitative diagnosis of spasticity and dystonia u=in CP. The study consists of face-to-face assessments of movement before, after, and one-month following the completion of the six-session game-based intervention. Children with spastic/dystonic cerebral palsy and typically developing children between the ages of 7 and 17 will be recruited for this study. The investigators anticipate to recruit a total of 68 participants, 34 with cerebral palsy and 34 typically developing. Both groups of children will be randomly allocated into an intervention or control group using a blocked randomization method. Movement outcomes will be examined for changes in quantitative and clinical measures in children with spastic/dystonic cerebral palsy and typically developing children to aid on the classification of movement disorders. Pair t-tests will be conducted on movement outcomes for both groups of children independently. Positive and negative results will be reported and addressed.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 7 and 17
* Have been diagnosed with dystonic or spastic/dystonic cerebral palsy, for the cerebral palsy groups, or have no neuromuscular conditions, for typically developing groups
* Have mild to no difficulty understanding conversations compared to others of the same age
* Communicates age appropriately or with some difficulty but a new listener can understand
* Have no uncorrected vision
* Have hearing without the need of a hearing aid
* Have no other neural, neuromuscular, or musculoskeletal conditions
* Participation in stable school and/or private physical or occupational therapy with a frequency no greater than two sessions per week, for cerebral palsy groups
* Have no changes in medication for the six months previous to enrollment in the study
* Be medically stable
* Have no other concurrent illness
* Have not received any Botox treatment within three months previous to the initiation of the study
* No use of cardiac pacemakers, hearing aids, or another electronic implanted device
* Absence of allergy to silver or skin adhesives
* Have never had seizures
* Have Manual Ability Classification System (MACS) score I-III

Exclusion Criteria:

* Not meeting ALL inclusion criteria

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Smoothness Index | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The smoothness index will be measured by analyzing the the integrated accelerometry signals of sensors placed on the upper limbs. Accelerometry data will be integrated to calculate the smoothness index on the velocity profile of the trajectories.
  The maximum value is 0, being the greatest level of smoothness that can be measured, and the minimum is minus infinity. A value closer to 0 is desired.

SECONDARY OUTCOMES:
Surface electromyography | Tested during the assessment sessions and on the first and last day of gameplay spanning over a 6 to 7 week period.
  Surface electromyography (sEMG) data will be collected during the execution of a first port de bras. The first port de bras will follow the format from the Royal Academy of Dance as demonstrated (Figure 1). Data will be analyzed changes in muscle activity patterns as a secondary outcome measure. The sEMG data will also be acquired during maximum voluntary efforts. For calibration of game-playing.
Forces and torques against force sensor during gampeplay and in robotic zero-force channel | Tested during the assessment sessions and on the first and last day of gameplay spanning over a 6 to 7 week period.
  This involves a force/torque sensor mounted in the end effector of the robot. A pre-determined zero-force path has been programmed by the research team to allow the robot to move through straight lines connected to five points on a vertical plane. The participants will hold a gripper mounted on the force transducer and attempt to move the end effector of the robot along the zero-force path. The force transducer will measure the forces exerted by the participant as they do so. Force and torque signals will be collected during all game-playing sessions. The calibration for game playing involves a maximum voluntary effort by the participant's dominant arm against the sensor mounted on a sturdy table. Participants will also be assessed with the force sensor in fourteen different directions at 30% ± 10% of the maximal voluntary effort across all directions.
Montreal Spasticity Rating Test (MSRT) | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The MSRT is a quantitative measure the onset of the stretch reflex that that correlates with clinical spasticity and shows good test re-test reliability
Dyskinesia Impairment Scale (DIS) | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The Dyskinesia Impairment Scale (DIS) measures the severity of dystonia and choreoathetosis when an individual is at rest or moving. It was found to show good to excellent reliability and validity. Scores range from 0 to 4 for both duration and amplitude of each criterion. A score of 0 most corresponds to movement of healthy people without movement disorders. The highest score possible score is 576 indicating the most server level of impairs,ent. There are two sub scales: Dystonia and Choreoathetosis that have a range of 0-288 each. The total score is obtained by addition of the two subscores.
Selective Control of the Upper Extremity Scale (SCUES) | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The Selective Control of the Upper Extremity Scale (SCUES) is a video-based tool to measure selective control of upper limb tasks. Psychometric analysis shows "comparable validity to other accepted video-based clinical assessment tools for the upper extremity in children with CP " with content validity ratio values indicating substantial agreement for most items. Scores are assigned for each assessed joint and can be rated as M3, M2, M1, or M0 with M3 representing normal selective motor control and M0 representing no selective motor control.
Quality of Upper Extremity Skills Test (QUEST) | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The QUEST is 36 items in length and measures upper limb movement, hand function, and cooperativeness in children with CP. It has been found to be reliable to assess children with CP between 18 months and 8 years of age, with increased reliability in children up to 12 years of age [30]. It has also been found to show adequate to excellent validity.
  Initial scores range from 50 to 100, which are then standardized to be between 0 and 100. The initial score is summed by scoring the ability to complete an item according to specification as 2 points, not being able to, not willing to, or not administerable as 1 point, and minus 1 point for abnormal movement in the posture section of the assessment. The standardized score is found by dividing the sum of scores for each section tested by the total number of sections tested.
Tardieu scale | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The Tardieu scale examines spasticity with quantified measures of the responses of stretch reflexes. This scale shows high test retest and poor to moderate inter-rater reliability; the Tardieu scale performs better than other similar measures, indicating it may be more reliable.
  Scores of quality of muscle reaction range from 0 to 5 with 0 being no resistance throughout passive movement and 5 being an immobile joint.
World Health Organization Disability Assessment Schedule 2 Children and Youth (WHODAS II - CY) | Tested during the assessment sessions spanning over a 6 to 7 week period.
  The WHODAS II - CY is a self-report 36 item document that assesses daily issues surrounding health conditions such as illnesses, injuries, and problems with mental health. In a validity study, it was found to show good reliability; however, limitations regarding options for those without significant disabilities were present.
  Each item can be scored from 1 to 5, with 1 indicating none and 5 indicating extreme or cannot do. Each item is scored, summed within the domain it is in, and the average is taken for each domain. The averages are summed and converted to a metric ranging from 0 to 100 where 0 indicates no disability and 100 indicating severe disability.
Qualitative Feedback Module | Tested during the assessment sessions spanning over a 6 to 7 week period.
  Multiple choice patient satisfaction questionnaire. Scores range from 0 to 5 for each item similar to the Wong-Baker FACES Pain Rating Scale with 0 indicating highest satisfaction and 5 indicating highest dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Citlali Lopez-Ortiz, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen D, Van Naarden Braun K, Doernberg NS, Maenner MJ, Arneson CL, Durkin MS, Benedict RE, Kirby RS, Wingate MS, Fitzgerald R, Yeargin-Allsopp M. Prevalence of cerebral palsy, co-occurring autism spectrum disorders, and motor functioning - Autism and Developmental Disabilities Monitoring Network, USA, 2008. Dev Med Child Neurol. 2014 Jan;56(1):59-65. doi: 10.1111/dmcn.12268. Epub 2013 Oct 1. PMID 24117446
- [Background] Paneth N. Establishing the diagnosis of cerebral palsy. Clin Obstet Gynecol. 2008 Dec;51(4):742-8. doi: 10.1097/GRF.0b013e318187081a. PMID 18981799
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Liptak GS. Health and well being of adults with cerebral palsy. Curr Opin Neurol. 2008 Apr;21(2):136-42. doi: 10.1097/WCO.0b013e3282f6a499. PMID 18317270
- [Background] Rice J, Skuza P, Baker F, Russo R, Fehlings D. Identification and measurement of dystonia in cerebral palsy. Dev Med Child Neurol. 2017 Dec;59(12):1249-1255. doi: 10.1111/dmcn.13502. Epub 2017 Aug 8. PMID 28786476
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Sanger TD. Arm trajectories in dyskinetic cerebral palsy have increased random variability. J Child Neurol. 2006 Jul;21(7):551-7. doi: 10.1177/08830738060210070201. PMID 16970842
- [Background] Sellier E, Platt MJ, Andersen GL, Krageloh-Mann I, De La Cruz J, Cans C; Surveillance of Cerebral Palsy Network. Decreasing prevalence in cerebral palsy: a multi-site European population-based study, 1980 to 2003. Dev Med Child Neurol. 2016 Jan;58(1):85-92. doi: 10.1111/dmcn.12865. Epub 2015 Aug 28. PMID 26330098
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Cramer SC, Sur M, Dobkin BH, O'Brien C, Sanger TD, Trojanowski JQ, Rumsey JM, Hicks R, Cameron J, Chen D, Chen WG, Cohen LG, deCharms C, Duffy CJ, Eden GF, Fetz EE, Filart R, Freund M, Grant SJ, Haber S, Kalivas PW, Kolb B, Kramer AF, Lynch M, Mayberg HS, McQuillen PS, Nitkin R, Pascual-Leone A, Reuter-Lorenz P, Schiff N, Sharma A, Shekim L, Stryker M, Sullivan EV, Vinogradov S. Harnessing neuroplasticity for clinical applications. Brain. 2011 Jun;134(Pt 6):1591-609. doi: 10.1093/brain/awr039. Epub 2011 Apr 10. PMID 21482550
- [Background] Sukal-Moulton T, Clancy T, Zhang LQ, Gaebler-Spira D. Clinical application of a robotic ankle training program for cerebral palsy compared to the research laboratory application: does it translate to practice? Arch Phys Med Rehabil. 2014 Aug;95(8):1433-40. doi: 10.1016/j.apmr.2014.04.010. Epub 2014 May 2. PMID 24792141
- [Background] Beveridge B, Feltracco D, Struyf J, Strauss E, Dang S, Phelan S, Wright FV, Gibson BE. "You gotta try it all": Parents' Experiences with Robotic Gait Training for their Children with Cerebral Palsy. Phys Occup Ther Pediatr. 2015;35(4):327-41. doi: 10.3109/01942638.2014.990547. Epub 2014 Dec 20. PMID 25529412
- [Background] Chen K, Ren Y, Gaebler-Spira D, Zhang LQ. Home-based tele-assisted robotic rehabilitation of joint impairments in children with cerebral palsy. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:5288-91. doi: 10.1109/EMBC.2014.6944819. PMID 25571187
- [Background] Krebs HI, Fasoli SE, Dipietro L, Fragala-Pinkham M, Hughes R, Stein J, Hogan N. Motor learning characterizes habilitation of children with hemiplegic cerebral palsy. Neurorehabil Neural Repair. 2012 Sep;26(7):855-60. doi: 10.1177/1545968311433427. Epub 2012 Feb 13. PMID 22331211
- [Background] Fasoli SE, Fragala-Pinkham M, Hughes R, Krebs HI, Hogan N, Stein J. Robotic therapy and botulinum toxin type A: a novel intervention approach for cerebral palsy. Am J Phys Med Rehabil. 2008 Dec;87(12):1022-5. doi: 10.1097/PHM.0b013e31817fb346. PMID 18617860
- [Background] Sanger TD, Kaiser J, Placek B. Reaching movements in childhood dystonia contain signal-dependent noise. J Child Neurol. 2005 Jun;20(6):489-96. doi: 10.1177/088307380502000604. PMID 15996397
- [Background] Jankovic J. Treatment of dystonia. Lancet Neurol. 2006 Oct;5(10):864-72. doi: 10.1016/S1474-4422(06)70574-9. PMID 16987733
- [Background] Damiano DL, DeJong SL. A systematic review of the effectiveness of treadmill training and body weight support in pediatric rehabilitation. J Neurol Phys Ther. 2009 Mar;33(1):27-44. doi: 10.1097/NPT.0b013e31819800e2. PMID 19265768
- [Background] Scianni A, Butler JM, Ada L, Teixeira-Salmela LF. Muscle strengthening is not effective in children and adolescents with cerebral palsy: a systematic review. Aust J Physiother. 2009;55(2):81-7. doi: 10.1016/s0004-9514(09)70037-6. PMID 19463078
- [Background] Deon LL, Gaebler-Spira D. Assessment and treatment of movement disorders in children with cerebral palsy. Orthop Clin North Am. 2010 Oct;41(4):507-17. doi: 10.1016/j.ocl.2010.06.001. PMID 20868881
- [Background] Bertucco M, Sanger TD. Current and emerging strategies for treatment of childhood dystonia. J Hand Ther. 2015 Apr-Jun;28(2):185-93; quiz 194. doi: 10.1016/j.jht.2014.11.002. Epub 2014 Nov 15. PMID 25835254
- [Background] Fehlings D, Brown L, Harvey A, Himmelmann K, Lin JP, Macintosh A, Mink JW, Monbaliu E, Rice J, Silver J, Switzer L, Walters I. Pharmacological and neurosurgical interventions for managing dystonia in cerebral palsy: a systematic review. Dev Med Child Neurol. 2018 Apr;60(4):356-366. doi: 10.1111/dmcn.13652. Epub 2018 Feb 6. PMID 29405267
- [Background] Bird BL, Cataldo MF. Experimental analysis of EMG feedback in treating dystonia. Ann Neurol. 1978 Apr;3(4):310-15. doi: 10.1002/ana.410030406. PMID 666271
- [Background] Neilson PD, McCaughey J. Self-regulation of spasm and spasticity in cerebral palsy. J Neurol Neurosurg Psychiatry. 1982 Apr;45(4):320-30. doi: 10.1136/jnnp.45.4.320. PMID 7077341
- [Background] Deepak KK, Behari M. Specific muscle EMG biofeedback for hand dystonia. Appl Psychophysiol Biofeedback. 1999 Dec;24(4):267-80. doi: 10.1023/a:1022239014808. PMID 10789003
- [Background] Lopez-Ortiz C, Gladden K, Deon L, Schmidt J, Girolami G, Gaebler-Spira D. Dance program for physical rehabilitation and participation in children with cerebral palsy. Arts Health. 2012 Feb 1;4(1):39-54. doi: 10.1080/17533015.2011.564193. Epub 2011 Jun 13. PMID 25431617
- [Background] Yamada K, Yamada Z, Nakazawa S, Matsuoka S. [Determination of FDP by staphylococcal clumping test and the significance of the method in consumption coagulopathy]. Rinsho Ketsueki. 1972 Jun;13(3):411-4. No abstract available. Japanese. PMID 4674971
- [Background] Jobin A, Levin MF. Regulation of stretch reflex threshold in elbow flexors in children with cerebral palsy: a new measure of spasticity. Dev Med Child Neurol. 2000 Aug;42(8):531-40. doi: 10.1017/s0012162200001018. PMID 10981931
- [Background] Monbaliu E, Ortibus E, De Cat J, Dan B, Heyrman L, Prinzie P, De Cock P, Feys H. The Dyskinesia Impairment Scale: a new instrument to measure dystonia and choreoathetosis in dyskinetic cerebral palsy. Dev Med Child Neurol. 2012 Mar;54(3):278-83. doi: 10.1111/j.1469-8749.2011.04209.x. PMID 22428172
- [Background] Stewart K, Harvey A, Johnston LM. A systematic review of scales to measure dystonia and choreoathetosis in children with dyskinetic cerebral palsy. Dev Med Child Neurol. 2017 Aug;59(8):786-795. doi: 10.1111/dmcn.13452. Epub 2017 May 9. PMID 28485494
- [Background] Wagner LV, Davids JR, Hardin JW. Selective Control of the Upper Extremity Scale: validation of a clinical assessment tool for children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2016 Jun;58(6):612-7. doi: 10.1111/dmcn.12949. Epub 2015 Nov 3. PMID 26526592
- [Background] Thorley M, Lannin N, Cusick A, Novak I, Boyd R. Reliability of the quality of upper extremity skills test for children with cerebral palsy aged 2 to 12 years. Phys Occup Ther Pediatr. 2012 Feb;32(1):4-21. doi: 10.3109/01942638.2011.602389. Epub 2011 Aug 15. PMID 21838618
- [Background] Law M, Cadman D, Rosenbaum P, Walter S, Russell D, DeMatteo C. Neurodevelopmental therapy and upper-extremity inhibitive casting for children with cerebral palsy. Dev Med Child Neurol. 1991 May;33(5):379-87. doi: 10.1111/j.1469-8749.1991.tb14897.x. PMID 2065824
- [Background] Klingels K, De Cock P, Desloovere K, Huenaerts C, Molenaers G, Van Nuland I, Huysmans A, Feys H. Comparison of the Melbourne Assessment of Unilateral Upper Limb Function and the Quality of Upper Extremity Skills Test in hemiplegic CP. Dev Med Child Neurol. 2008 Dec;50(12):904-9. doi: 10.1111/j.1469-8749.2008.03123.x. Epub 2008 Sep 20. PMID 18811701
- [Background] Mehrholz J, Wagner K, Meissner D, Grundmann K, Zange C, Koch R, Pohl M. Reliability of the Modified Tardieu Scale and the Modified Ashworth Scale in adult patients with severe brain injury: a comparison study. Clin Rehabil. 2005 Oct;19(7):751-9. doi: 10.1191/0269215505cr889oa. PMID 16250194
- [Background] Wolf AC, Tate RL, Lannin NA, Middleton J, Lane-Brown A, Cameron ID. The World Health Organization Disability Assessment Scale, WHODAS II: reliability and validity in the measurement of activity and participation in a spinal cord injury population. J Rehabil Med. 2012 Sep;44(9):747-55. doi: 10.2340/16501977-1016. PMID 22854805
- [Background] Young SJ, van Doornik J, Sanger TD. Finger muscle control in children with dystonia. Mov Disord. 2011 Jun;26(7):1290-6. doi: 10.1002/mds.23534. Epub 2011 Mar 29. PMID 21449015
- [Background] Frascarelli F, Masia L, Di Rosa G, Cappa P, Petrarca M, Castelli E, Krebs HI. The impact of robotic rehabilitation in children with acquired or congenital movement disorders. Eur J Phys Rehabil Med. 2009 Mar;45(1):135-41. PMID 19293759
- [Background] Weightman A, Preston N, Levesley M, Holt R, Mon-Williams M, Clarke M, Cozens AJ, Bhakta B. Home based computer-assisted upper limb exercise for young children with cerebral palsy: a feasibility study investigating impact on motor control and functional outcome. J Rehabil Med. 2011 Mar;43(4):359-63. doi: 10.2340/16501977-0679. PMID 21347508
- [Background] Chen YP, Howard AM. Effects of robotic therapy on upper-extremity function in children with cerebral palsy: A systematic review. Dev Neurorehabil. 2016;19(1):64-71. doi: 10.3109/17518423.2014.899648. Epub 2014 Apr 11. PMID 24724587
- [Background] Gilliaux M, Renders A, Dispa D, Holvoet D, Sapin J, Dehez B, Detrembleur C, Lejeune TM, Stoquart G. Upper limb robot-assisted therapy in cerebral palsy: a single-blind randomized controlled trial. Neurorehabil Neural Repair. 2015 Feb;29(2):183-92. doi: 10.1177/1545968314541172. Epub 2014 Jul 11. PMID 25015650
- [Background] Tong LZ, Ong HT, Tan JX, Lin J, Burdet E, Ge SS, Teo CL. Pediatric rehabilitation with the reachMAN's modular handle. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:3933-6. doi: 10.1109/EMBC.2015.7319254. PMID 26737154
- [Background] Preston N, Weightman A, Gallagher J, Holt R, Clarke M, Mon-Williams M, Levesley M, Bhakta B. Feasibility of school-based computer-assisted robotic gaming technology for upper limb rehabilitation of children with cerebral palsy. Disabil Rehabil Assist Technol. 2016;11(4):281-8. doi: 10.3109/17483107.2014.932020. Epub 2014 Jun 25. PMID 24964205
- [Background] Kluzik J, Fetters L, Coryell J. Quantification of control: a preliminary study of effects of neurodevelopmental treatment on reaching in children with spastic cerebral palsy. Phys Ther. 1990 Feb;70(2):65-76; discussion 76-8. doi: 10.1093/ptj/70.2.65. PMID 2296614
- [Background] Volman MJ, Wijnroks A, Vermeer A. Effect of task context on reaching performance in children with spastic hemiparesis. Clin Rehabil. 2002 Sep;16(6):684-92. doi: 10.1191/0269215502cr540oa. PMID 12392345
- [Background] Johansson AM, Domellof E, Ronnqvist L. Short- and long-term effects of synchronized metronome training in children with hemiplegic cerebral palsy: a two case study. Dev Neurorehabil. 2012;15(2):160-9. doi: 10.3109/17518423.2011.635608. Epub 2012 Feb 1. PMID 22296344
- [Background] Lebiedowska MK, Gaebler-Spira D, Burns RS, Fisk JR. Biomechanic characteristics of patients with spastic and dystonic hypertonia in cerebral palsy. Arch Phys Med Rehabil. 2004 Jun;85(6):875-80. doi: 10.1016/j.apmr.2003.06.032. PMID 15179639
- [Background] Gordon LM, Keller JL, Stashinko EE, Hoon AH, Bastian AJ. Can spasticity and dystonia be independently measured in cerebral palsy? Pediatr Neurol. 2006 Dec;35(6):375-81. doi: 10.1016/j.pediatrneurol.2006.06.015. PMID 17138005
- [Background] Kim Y, Bulea TC, Damiano DL. Children With Cerebral Palsy Have Greater Stride-to-Stride Variability of Muscle Synergies During Gait Than Typically Developing Children: Implications for Motor Control Complexity. Neurorehabil Neural Repair. 2018 Sep;32(9):834-844. doi: 10.1177/1545968318796333. PMID 30223739
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773
- [Background] Tedroff K, Knutson LM, Soderberg GL. Synergistic muscle activation during maximum voluntary contractions in children with and without spastic cerebral palsy. Dev Med Child Neurol. 2006 Oct;48(10):789-96. doi: 10.1017/S0012162206001721. PMID 16978457
- [Background] Quartarone A, Rizzo V, Morgante F. Clinical features of dystonia: a pathophysiological revisitation. Curr Opin Neurol. 2008 Aug;21(4):484-90. doi: 10.1097/WCO.0b013e328307bf07. PMID 18607211
- [Background] Mink JW. Special concerns in defining, studying, and treating dystonia in children. Mov Disord. 2013 Jun 15;28(7):921-5. doi: 10.1002/mds.25548. PMID 23893449
- [Derived] McNish RN, Chembrammel P, Speidel NC, Lin JJ, Lopez-Ortiz C. Rehabilitation for Children With Dystonic Cerebral Palsy Using Haptic Feedback in Virtual Reality: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 14;8(1):e11470. doi: 10.2196/11470. PMID 31344678